CLINICAL TRIAL: NCT03013881
Title: Open-label, Two-part, Dose-escalation and Comparative Pharmacokinetics Study of UB-921 in Healthy Male Volunteers
Brief Title: A Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of UB-921 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: United BioPharma (Industry)
Collaborators: Tri-Service General Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UBP-A103-HER2
Record Dates: First submitted 2017-01-02; First posted 2017-01-09 (Estimated); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Breast Neoplasm
Keywords: UB-921; anti-HER2 monoclonal antibody; breast neoplasm; breast cancer; Herceptin; Trastuzumab; HER2
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- UB-921 2 mg/kg (Main-study) (Experimental): Intravenous infusion
  Interventions: Biological: UB-921
- UB-921 6 mg/kg (Main-study) (Experimental): Intravenous infusion
  Interventions: Biological: UB-921
- UB-921 8 mg/kg (Main-study) (Experimental): Intravenous infusion
  Interventions: Biological: UB-921
- UB-921 6 mg/kg (Sub-study) (Experimental): Intravenous infusion
  Interventions: Biological: UB-921
- Herceptin 6 mg/kg (Sub-study) (Active Comparator): Intravenous infusion
  Interventions: Biological: Herceptin

INTERVENTIONS:
Biological: UB-921 — 150 mg/vial
  Arms: UB-921 2 mg/kg (Main-study); UB-921 6 mg/kg (Main-study); UB-921 6 mg/kg (Sub-study); UB-921 8 mg/kg (Main-study)
Biological: Herceptin — 440 mg/vial
  Arms: Herceptin 6 mg/kg (Sub-study)

SUMMARY:
The purpose of the study is to evaluate the safety, tolerability, and pharmacokinetics of escalating single-dose of UB-921 in healthy male volunteers.

DETAILED DESCRIPTION:
This is an open-label, two-part, dose-escalation and comparative pharmacokinetics study of UB-921 in healthy male volunteers. There will be two parts: dose escalation study (Main Study) and comparative pharmacokinetics study (Sub-study).

ELIGIBILITY:
Inclusion Criteria:

* Total body weight ≧50 kg (110 lbs)
* No clinically relevant abnormalities
* To agree on using birth control barrier (eg. male condom) during the entire study period.
* Signing the written informed consent form

Exclusion Criteria:

* Previous exposure to chimeric, humanized or human monoclonal antibody, whether licensed or investigational
* A history of drug abuse or heavy drinking.
* Blood donation over 250 mL within 90 days prior to the screening
* Not in the condition to participate in this study considered by investigator(s)

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2018-10-08 (Actual); Study Completion 2019-04-02 (Actual)

PRIMARY OUTCOMES:
Adverse event incidence | 63 days
  from the baseline to the end of study visit

CONTACTS AND LOCATIONS:
Overall Officials: Hsiang-Cheng Chen, Principal Investigator — Tri-Service General Hospital
Locations (1):
- Prime site, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No